CLINICAL TRIAL: NCT05667922
Title: Development and Validation of a Prognostic Model for Idiopathic Membranous Nephropathy Treated With Tacrolimus
Brief Title: Prognostic Model of TAC in the Treatment of MN
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Zunsong Wang, Principal Investigator, Qianfoshan Hospital
Other Study IDs: IMN-TAC
Record Dates: First submitted 2022-12-07; First posted 2022-12-29 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Idiopathic Membranous Nephropathy
MeSH Terms: conditions — Glomerulonephritis, Membranous | interventions — Tacrolimus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Remission
  Interventions: Drug: Tacrolimus
- Non-remission
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — 0.05-0.10mg/kg/d, twice orally, with an interval of 12h. The drug valley concentration is 5-10ng/ml, which will be gradually reduced to a low dose after it is effective.

SUMMARY:
The goal of this observational study is to explore the factors that can predict the prognosis difference in patients with idiopathic membranous nephropathy (IMN) under the treatment of tacrolimus. The main questions it aims to answer are:

* to explore the factors that can predict the prognosis difference in patients with IMN under the treatment of tacrolimus
* to establish a clinical prediction model and verify it to provide a reference for the early Participants will receive standard the treatment of tacrolimus treatment and will then be divided into remission and non remission groups based on the treatment effect after the standard treatment cycle. Blood, urine, and fecal samples were collected from patients to explore possible factors influencing treatment efficacy.

Researchers will compare [remission group and non-remission group] to see if the gut microbiota and its metabolites are factors that influence the efficacy of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years, the patient was diagnosed as idiopathic membranous nephropathy or anti phospholipase A2 receptor (PLA2R) antibody positive by renal puncture biopsy, and the clinical data were complete;
2. According to the Kidney Disease: Improving Global Outcomes (KDIGO) guidelines in 2020, it conforms to the medium and high risks in the risk level of progression of renal function loss.
3. In general, they are in good condition, have a good understanding of their own conditions and physical conditions, have self-awareness, and can communicate well with others;
4. Volunteer to participate in the study, understand the significance of this experiment and the indicators to be measured, and sign the informed consent form.

Exclusion Criteria:

1. There are factors causing secondary membranous nephropathy, such as immune diseases (systemic lupus erythematosus), tumors/infections (viral hepatitis), drugs or toxins;
2. At the same time, immunoglobulin A nephropathy (IgAN), interstitial nephritis, acute nephritis and other renal pathological types were combined;
3. The medication was not standardized during the treatment process, accompanied by serious infection, acute renal injury and other complications, and serious cardiovascular, cerebrovascular, digestive and blood system diseases;
4. During follow-up, the patient cannot actively cooperate or accurately understand and express.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with idiopathic membranous nephropathy diagnosed at age 18-75 years
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Remission | 6 months
  1. None-Remission of the State of MN: 1)24-hour urin protein (24-h UP)>3.5 g, or 24-h UP<50% lower than the baseline, or serum creatinine increased by 50% compared with the baseline; 2) Renal function progress: Compared with the initial examination, estimated glomerular filtration rate (eGFR) progress is greater than or equal to 30%; 3) End stage renal disease: eGFR<15ml/min, or renal replacement therapy.
  2. Partial Remission of the State of MN: 24-h UP is 0.5-3.5 g, and 24-h UP is more than 50% lower than the baseline, serum creatinine is normal, and plasma albumin is ≥ 30 g.
  3. Complete remission of the State of MN: 24-h UP<0.5g, serum creatinine normal, plasma albumin ≥ 35g.

IPD SHARING:
Plan to Share IPD: No